CLINICAL TRIAL: NCT05534880
Title: Analysis of Cortical Activity in Individuals With Cybersickness Under the Influence of Multi-sensory Conditions in Virtual Reality: a Randomized Crossover Study
Brief Title: Cybersickness in Different Multisensory Conditions in Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Marcos Junio da Costa Silva, Undegraduate, Federal University of Piaui
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UFDPar
Record Dates: First submitted 2022-09-04; First posted 2022-09-10 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Cybersickness; Reduced Sensation
Keywords: cybersickness; virtual reality; binaural beats; electroencephalography
MeSH Terms: conditions — Hypesthesia

STUDY DESIGN:
Intervention Model Description: The study will be a double-blind randomized controlled clinical trial, with university students of both sexes in the city of Parnaíba - PI, volunteers who present cybersickness will be evaluated, those who meet the admission criteria will be randomized and allocated and will be immersed in three conditions, in these conditions the volunteers will be immersed in VR to induce symptoms, where bimodal conditions will be analyzed and compared to analyze the variable electrophysiological activity and the influence of multisensory conditions.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will not be aware of the intention of each of the immersion conditions, and will be randomized through a program for each of the conditions, by a researcher external to the research, and sorted through an opaque envelope, the participants and the researcher, not will know in which condition they will be allocated, only on the day of the draw, each participant will be allocated in the condition and the researcher will not be aware of which condition the participant will be immersed in (condition 01 - video only) or (condition 02 - video associated with binaural beat) .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Active Comparator): Condition 01 - the participants will be induced to CS, they will be immersed in a roller coaster simulation video, lasting 10 minutes, there will be 03 sessions on alternate days with a 24-hour interval between each session, before and after each session will be applied the SSQ questionnaire subjective assessment and EEG objective assessment.
  Interventions: Other: Binaural beats
- Virtual reality and binaural beats (Experimental): Condition 02 - the participants will be induced to CS, they will be immersed in a roller coaster simulation video associated with audio with binaural beat, lasting 10 minutes, there will be 03 sessions on alternate days with a 24-hour interval between each session, before and after each session, the SSQ subjective assessment questionnaire and the objective assessment EEG will be applied.
  Interventions: Other: Binaural beats

INTERVENTIONS:
Other: Binaural beats — Condition 02- will be used binaural beats, since they are referred through studies with the ability to drive neural oscillations in the beat frequency through differential hemispheric synchronization frequencies, it is expected that a neuromodulation and repercussion of the symptomatological reduction of CS.

SUMMARY:
Cybersickness (CS) is characterized as a type of visually induced motion sickness, similar to traditional motion sickness, with specific clinical presentations such as dizziness, eyestrain, oculomotor disorders, blurred vision and spatial disorientation. It can be triggered when experiencing virtual reality (VR), and it affects approximately 20% to 80% of individuals who use these resources. Furthermore, the underlying mechanisms of CS are not fully understood and the use of virtual environments that have become increasingly recurrent in several sectors deserves attention, as VR is becoming commonplace in methods and techniques of assessment, diagnosis and treatment. Objective: to analyze cortical electrophysiological activity using electroencephalography (EEG) in individuals with SC, under the influence of different audiovisual conditions. Methodology: The study is a double-blind randomized controlled clinical trial, the sample for survey satisfaction N= 10 participants, the public were university students from the Universidade Federal do Delta Parnaíba (UFDPar) of both sexes, aged between 18 to 28 years, those who agreed, underwent screening, those who met the criteria and fit, were randomized and allocated to one each of 02 conditions, (C1 - video only) and (C2 - associated with binaural audio), three times in each condition, with a duration of 10 minutes of immersion, with evaluation (pre) before (post) with QEEG and Sickness Questionnaire (SSQ), exposure to virtual content was on regular alternate days, with a 24-hour interval between each virtual exposure, at the end of each condition, there will be a 14-day washout and crossover between the conditions. The study will be carried out under all cleaning and prevention care in the fight against the Covid-19 pandemic, data collection will be at the Brain Mapping and Functionality Laboratory (LAMCEF) of the Federal University of Delta do Parnaíba, Piauí, Brazil. Results: The condition with binaural stimulation is expected to promote neuromodulation and reduction of CS symptoms, compared to the control condition.

DETAILED DESCRIPTION:
Objectives

General Objective

• Analyze whether the electrophysiological activity of the brain cortex of individuals with cybersickness undergoes neuromodulation through binaural stimuli;

Specific Objectives

* Investigate whether stimulation by binaural beats can mitigate the degree of symptoms through the SSQ;
* Compare whether there is a significant reduction in Sickness Questionare Simulator scores between conditions;
* Check if there is a difference in absolute power in the Delta band frequency of the parietal and frontal regions between the conditions;

Hypothesis

Our hypothesis is that the condition associated with binaural beats can promote neuromodulation in the electrophysiological activity of the brain cortex, altering the rhythms of brain wave frequencies, which can reduce sensory conflict in cybersickness, through wave entrainment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have normal or corrected to normal vision
* Participant must have a history of visually induced motion sickness

Exclusion Criteria:

* Cannot present vestibular disorders
* Claustrophobia
* Epileptic seizures
* Musculoskeletal disorders
* psychoactive drug use
* Neurological disorders
* Considerable hearing loss

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
analysis of electrophysiological activity | In pre-intervention procedures, the baseline cortical electroencephalography will be analyzed for 5 minutes. After immersion, the same procedures will be performed
  Analisys of absolute power of the Delta band frequencies of the frontal and temporand regions of the brain.

SECONDARY OUTCOMES:
Analysis of symptoms through the SSQ questionnaire | In the pre-intervention procedures, before the cortical analysis, the SSQ instrument will be applied, and immediately after each session, the subjective assessment instrument will be applied
  Simulator Sickness Questionnaire (SSQ) is a widely used tool to assess the subjective severity of symptoms of simulator illness and cybersickness. It consists of 16 items, on a four-point scale (from 'none' to 'severe').

CONTACTS AND LOCATIONS:
Overall Officials: Victor H. Bastos, Ph. D, Principal Investigator — Federal University of the Parnaiba Delta
Locations (2):
- Brazil (2):
  - Federal University of the Delta Parnaíba, Parnaíba, Piauí
  - Federal University of the Parnaiba Delta, Parnaíba, Piauí

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Dissociating vestibular and somatosensory contributions to spatial orientation — https://pubmed.ncbi.nlm.nih.gov/27075537/
- See also: The Potential of Immersive Virtual Reality for Cognitive Training in Elderly — https://pubmed.ncbi.nlm.nih.gov/32906122/
- See also: Simulator Sickness Questionnaire: tradução e adaptação transcultural — https://www.scielo.br/j/jbpsiq/a/trfYrY8LfWzmpwh7Wqn9Cvr/?lang=pt#:~:text=O%20Simulator%20Sickness%20Questionnaire%20(SSQ,o%20n%C3%ADvel%20de%20cybersickness14.
- See also: A Failure to Enhance EEG Power and Emotional Arousal — https://pubmed.ncbi.nlm.nih.gov/29187819/
- See also: The role of virtual reality in improving motor performance as revealed by EEG: a randomized clinical trial — https://pubmed.ncbi.nlm.nih.gov/28592282/
- See also: Humans integrate visual and haptic information in a statistically optimal fashion — https://pubmed.ncbi.nlm.nih.gov/28592282/
- See also: The Effects of Binaural and Monoaural Beat Stimulation on Cognitive Functioning in Subjects with Different Levels of Emotionality — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7204407/
- See also: Vestibular-somatosensory interactions: A mechanism in search of a function? — https://pubmed.ncbi.nlm.nih.gov/26595956/
- See also: Too Real to Be Virtual: Autonomic and EEG Responses to Extreme Stress Scenarios in Virtual Reality — https://pubmed.ncbi.nlm.nih.gov/32256856/
- See also: Efficacy of binaural auditory beats in cognition, anxiety, and pain perception: a meta-analysis — https://pubmed.ncbi.nlm.nih.gov/30073406/
- See also: Multisensory integration in self motion perception. Multisensory Research — https://brill.com/view/journals/msr/29/6-7/article-p525_2.xml
- See also: Cybersickness: A multisensory integration perspective — https://pubmed.ncbi.nlm.nih.gov/31264611/
- See also: Vection in virtual reality modulates vestibular-evoked myogenic potentials — https://pubmed.ncbi.nlm.nih.gov/31233640/
- See also: Binaural interaction of a beating frequency following response — https://pubmed.ncbi.nlm.nih.gov/7352918/
- See also: A meta-analysis of the virtual reality problem: Unequal effects of virtual reality sickness across individual differences — https://link.springer.com/article/10.1007/s10055-021-00524-3